CLINICAL TRIAL: NCT02166697
Title: Candesartan Cilexetil Tablets Specified Drug-use Survey "Hypertension: Survey on Patients With Metabolic Syndrome"
Brief Title: Blopress Tablets Specified Drug-use Survey "Hypertension: Survey on Patients With Metabolic Syndrome"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 460-015; JapicCTI-142567 (Registry Identifier: JapicCTI); JapicCTI-R160847 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Hypertension
Keywords: Pharmacological therapy
MeSH Terms: conditions — Hypertension | interventions — candesartan cilexetil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Oral administration of 4-8 mg of candesartan cilexetil: Oral administration of 4-8 milligram (mg) of candesartan cilexetil once daily (increased up to 12 mg, as necessary)
  Interventions: Drug: candesartan cilexetil

INTERVENTIONS:
Drug: candesartan cilexetil — candesartan cilexetil tablets
  Other Names: Blopress Tablets

SUMMARY:
The purpose of this survey is designed to investigate the treatment status of hypertensive patient with metabolic syndrome-related risk factors treated with candesartan cilexetil tablets (Blopress Tablets), as well as to assess relationships between risk factors (example, visceral fat accumulation) and the incidence of cerebrovascular/cardiovascular events in an exploratory manner.

DETAILED DESCRIPTION:
This survey was designed to investigate the treatment status of hypertensive patients with metabolic syndrome-related risk factors treated with candesartan cilexetil tablets (Blopress Tablets), as well as to assess relationships between risk factors (example, visceral fat accumulation) and the incidence of cerebrovascular/cardiovascular events in an exploratory manner.

For adults, 4-8 mg of candesartan cilexetil is typically administered orally once daily. The dose is increased up to 12 mg, as necessary. For patients with complications of renal damage, however, administration of candesartan cilexetil should be started at 2 mg once daily, and, as necessary, the dose increased up to 8 mg.

ELIGIBILITY:
Inclusion Criteria: Hypertensive patients with at least one of the following risk factors:

* Waist circumference greater than or equal to (≥) 85 centimeter (cm) for male and ≥ 90 cm for female
* Fasting triglyceride level ≥ 150 milligram per deciliter (mg/dL)
* High-density lipoprotein (HDL) cholesterol level less than (<) 40 mg/dL
* Fasting blood glucose level ≥ 110 mg/dL
* Body-mass index (BMI) ≥ 25.0 * Patients currently taking medications for hypertriglyceridemia, hypo-HDL-cholesterolemia, or diabetes mellitus are also regarded as meeting the criteria for inclusion in the surveillance

Exclusion Criteria: Hypertensive patients who meet all of the following conditions ([1] to [3]):

1. Patients receiving continuous therapy with Blopress Tablets
2. Patients aged < 20 years or ≥ 75 years
3. Patients with a history of cerebrovascular or coronary artery disease within 6 months before the start of the surveillance

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertension
Sampling Method: Non-Probability Sample
Enrollment: 14151 (Actual)
Dates: Start 2006-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Postmarketing Group Manager, Study Chair — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1,126 investigative sites in Japan from 7 June 2006 to 30 November 2010.
Pre-assignment Details: Participants with a historical diagnosis of hypertension with metabolic syndrome-related risk factors were observed in a single treatment group to receive candesartan cilexetil 4 milligrams (mg).
Groups:
- Candesartan Cilexetil: Candesartan cilexetil 4 mg, tablet, orally, once daily for up to 3 years.
Period: Overall Study
Arm/Group | Candesartan Cilexetil
Started | 14151
Completed | 13804
Not Completed | 347
Not completed — Protocol Violation | 347

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were enrolled and completed the study.
Arm/Group | Candesartan Cilexetil
Number analyzed (Participants) | 13804
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6087
  Male | 7717
Initial Daily Dose of Blopress [Number; unit: Participants]
  Less than (<) 4 mg | 214
  4 mg | 3934
  6 mg | 38
  8 mg | 8505
  10 mg | 1
  12 mg | 1104
  Greater than (>) 12 mg | 8
Blood Pressure [Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)]
  Systolic Blood Pressure | 156.2 (17.9)
  Diastolic Blood Pressure | 90.2 (12.6)
Pulse Rate [Mean (Standard Deviation); unit: Pulse per minute] | 73.9 (10.7)
Height [Mean (Standard Deviation); unit: Centimeter (cm)] | 160.28 (9.42)
Weight [Mean (Standard Deviation); unit: Kilogram (Kg)] | 68.07 (12.84)
Body Mass Index [Mean (Standard Deviation); unit: Kilogram per square meter (kg/m^2)] | 26.40 (3.84)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 90.56 (9.76)
Fasting Triglycerides [Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)] | 166.1 (101.6)
High Density Lipoprotein (HDL) Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 55.0 (15.2)
Fasting Blood Glucose [Mean (Standard Deviation); unit: mg/dL] | 118.4 (41.9)
Glycated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: Hemoglobin Percent] — It is reported as per National Glycohemoglobin Standardization Program (NGSP) value.
  Hemoglobin Percent | 6.46 (1.36)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 212.1 (37.7)
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.76 (0.29)
Urinary Protein [Number; unit: Participants] — Protein dipstick grading was used to analyze concentration of urinary protein.
  Participants
    0 mg/dL | 8365
    15-30mg/dL | 1005
    30-300mg/dL | 836
    100-300mg/dL | 440
    300-1000mg/dL | 185
    Unknown | 2973
Urinary Sugar [Number; unit: Participants]
  0 mg/dL | 8907
  100 mg/dL | 406
  250 mg/dL | 596
  500 mg/dL | 330
  1000 mg/dL | 566
  Unknown | 2999
Microalbumin in Urine [Mean (Standard Deviation); unit: Milligram per day (mg/day)] | 158.5 (653.6)
Insulin [Mean (Standard Deviation); unit: mcU/mL] — mcU/mL stands for micro international units per milliliter.
  mcU/mL | 11.09 (11.38)
Apoprotein A [Mean (Standard Deviation); unit: mg/dL] | 145.4 (24.5)
Apoprotein B [Mean (Standard Deviation); unit: mg/dL] | 104.1 (27.5)
Adiponectin [Mean (Standard Deviation); unit: Microgram per milliliter (mcg/mL)] | 5.80 (6.92)
Leptin [Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)] | 9.20 (8.24)
Smoking Status [Number; unit: Participants]
  Non Smoker | 10823
  Smoker | 2981
Alcohol Consumption [Number; unit: Participants]
  Alcohol Non-Consumer | 8265
  Alcohol Consumer | 5539
Predisposition to Hypersensitivity [Number; unit: Participants]
  Had no Predisposition to Hypersensitivity | 12259
  Had Predisposition to Hypersensitivity | 691
  Unknown | 854
Medical History [Number; unit: Participants]
  Did not Have Medical History | 3833
  Have Medical History | 9835
  Unknown | 136
Breakdown of Medical History [Number; unit: Participants] — Participants may be represented in more than 1 category.
  Participants
    Cerebral Infarction | 593
    Cerebral Hemorrhage | 63
    Subarachnoid Hemorrhage | 22
    Myocardial Infarction | 153
    Cardiac Failure | 121
    Angina Pectoris | 463
    Diabetes Mellitus | 4755
    Hyperlipidemia | 7841
    Other Cerebrovascular/Cardiovascular Diseases | 615
    Diabetic Retinopathy | 3
    Renal Dialysis | 0
    Atrial fibrillation | 257
Consumption of Concomitant Antihypertensive Medications [Number; unit: Participants]
  Had no Consumption | 8006
  Had Consumption | 5798
Breakdown of Concomitant Antihypertensive Medications [Number; unit: Participants] — Participants may be represented in more than 1 category.
  Participants
    Diuretics | 705
    Alpha-Blockers | 323
    Alpha-Beta or Beta-Blockers | 867
    Calcium Blockers | 4886
    Angiotensin Converting Enzyme (ACE) Inhibitors | 262
    Angiotensin2ReceptorBlockers(other than Blopress) | 131
    Other | 69
Consumption of Concomitant Antidiabetic Medications [Number; unit: Participants]
  Had no consumption | 10494
  Had Consumption | 3310
Breakdown of Concomitant Antidiabetic Medications [Number; unit: Participants] — Participants may be represented in more than 1 category.
  Participants
    Alpha-Glucosidase Inhibitor | 1127
    Insulin Sensitizers | 1077
    Sulfonylurea Drugs | 1728
    Short Acting Insulin Secretagogues | 306
    Biguanides | 686
    Insulin | 364
    Other | 44
Consumption of Concomitant Antihyperlipidemic Drugs [Number; unit: Participants]
  Had no Consumption | 9112
  Had Consumption | 4692
Breakdown of Concomitant Antihyperlipidemic Drugs [Number; unit: Participants] — Participants may be represented in more than 1 category.
  Participants
    Statins | 3784
    Fibrates | 730
    Eicosapentaenoic Acid | 230
    Other | 122
Consumption of Other Concomitant Medications [Number; unit: Participants]
  Had no Consumption | 9110
  Had Consumption | 4694
Breakdown of Other Concomitant Medication [Number; unit: Participants] — Participants may be represented in more than 1 category.
  Participants
    Antithrombotic Drugs | 1322
    Antigout Drugs or Antihyperuricemic Drugs | 903
    Other | 3005
Pulse Wave Velocity [Mean (Standard Deviation); unit: Centimeter per second (cm/s)] — Pulse wave velocity (PWV) is a measure of arterial stiffness, or the rate at which pressure waves move down the vessel.
  Centimeter per second (cm/s) | 1713.8 (523.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Adverse Drug Reactions (ADR)
Description: ADR are defined as adverse events (AEs) which are in the investigator's opinion of causal relationship to the study treatment. AEs are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug.
Time Frame: Baseline up to 3 years
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Measure: Number; unit: Participants
Arm/Group | Candesartan Cilexetil
Number analyzed (Participants) | 13804
Participants | 230

2. Primary Outcome: Number of Participants Reporting One or More Serious Adverse Drug Reactions (SADR)
Description: SADR are defined as serious adverse events (SAEs) which are in the investigator's opinion of causal relationship to the study treatment. SADR was an ADR resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to 3 years
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Measure: Number; unit: Participants
Arm/Group | Candesartan Cilexetil
Number analyzed (Participants) | 13804
Participants | 320

3. Secondary Outcome: Incidence of Cerebrovascular/Cardiovascular Events
Description: Cerebrovascular/cardiovascular events reported to be associated with Blopress were reported. The composite events classified under primary major adverse cardiac Events (MACE) 1 and primary MACE2 were defined as: MACE1: sudden death, cerebral hemorrhage, cerebral infarction, subarachnoid hemorrhage, and acute myocardial infarction; MACE2: MACE1 + hospitalization for cardiac failure and intervention/hospitalization for angina pectoris. Renal events include (transition to dialysis + renal transplant).
Time Frame: Baseline up to 3 years
Population: The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available.
Measure: Number; unit: Number of events per 1,000 person-years
Arm/Group | Candesartan Cilexetil
Number analyzed (Participants) | 13804
Number of events per 1,000 person-years
  Sudden Death | 0.24
  Cerebral Hemorrhage | 0.57
  Cerebral Infarction | 2.34
  Subarachnoid Hemorrhage | 0.15
  Acute Myocardial Infarction | 0.99
  Hospitalization for Heart Failure | 0.27
  Intervention/Hospitalization for Angina Pectoris | 1.74
  Atrial Fibrillation | 1.35
  Transition to Dialysis | 0.30
  Renal Transplant | 0.00
  Dissecting Aortic Aneurysm | 0.06
  Diabetic Retinopathy | 0.15
  New-Onset Diabetes | 4.35
  Primary MACE | 4.29
  Primary MACE 2 | 6.29
  Renal Events | 0.30

4. Secondary Outcome: Incidence of Cerebrovascular/Cardiovascular Events Affected by Underlying Risk Factors of Obesity, Blood Glucose Abnormalities, or Lipid Abnormalities
Description: Participants reporting cerebrovascular/cardiovascular events who had either obesity, blood glucose abnormalities, or lipid abnormalities as any one of the underlying risk factors associated with Blopress at the time of enrollment were reported.The composite events classified under primary MACE1 and primary MACE2 were defined as: MACE1: sudden death, cerebral hemorrhage, cerebral infarction, subarachnoid hemorrhage, and acute myocardial infarction; MACE2: MACE1 + hospitalization for cardiac failure and intervention/hospitalization for angina pectoris. Renal events include (transition to dialysis + renal transplant).
Time Frame: Baseline up to 3 years
Population: as for outcome 3
Measure: Number; unit: Number of events/1,000 person-years
Arm/Group | Candesartan Cilexetil
Number analyzed (Participants) | 4056
Number of events/1,000 person-years
  Sudden Death | 0.21
  Cerebral Hemorrhage | 0.41
  Cerebral Infarction | 1.55
  Subarachnoid Hemorrhage | 0.10
  Acute Myocardial Infarction | 0.62
  Hospitalization for Heart Failure | 0.10
  Intervention/Hospitalization for Angina Pectoris | 1.45
  Atrial Fibrillation | 0.62
  Transition to Dialysis | 0.31
  Renal Transplant | 0.00
  Dissecting Aortic Aneurysm | 0.00
  Diabetic Retinopathy | 0.10
  New-Onset Diabetes | 3.32
  Primary MACE | 2.90
  Primary MACE 2 | 4.45
  Renal Events | 0.31

5. Secondary Outcome: Incidence of Cerebrovascular/Cardiovascular Events Affected by Underlying Risk Factors of Obesity + Blood Glucose Abnormalities, Obesity + Lipid Abnormalities, or Blood Glucose Abnormalities + Lipid Abnormalities
Description: Participants reporting cerebrovascular/cardiovascular events who had multiple underlying risk factors which included either obesity + blood glucose abnormalities, obesity + lipid abnormalities OR blood glucose + lipid abnormalities associated with Blopress at the time of enrollment were reported. The composite events classified under primary MACE1 and primary MACE2 were defined as: MACE1: sudden death, cerebral hemorrhage, cerebral infarction, subarachnoid hemorrhage, and acute myocardial infarction; MACE2: MACE1 + hospitalization for cardiac failure and intervention/hospitalization for angina pectoris. Renal events include (transition to dialysis + renal transplant).
Time Frame: Baseline up to 3 years
Population: as for outcome 3
Measure: Number; unit: Number of events/1,000 person-years
Arm/Group | Candesartan Cilexetil
Number analyzed (Participants) | 6216
Number of events/1,000 person-years
  Sudden Death | 0.20
  Cerebral Hemorrhage | 0.53
  Cerebral Infarction | 2.19
  Subarachnoid Hemorrhage | 0.13
  Acute Myocardial Infarction | 1.06
  Hospitalization for heart Failure | 0.33
  Intervention/Hospitalization for Angina Pectoris | 1.33
  Atrial Fibrillation | 1.46
  Transition to Dialysis | 0.07
  Renal Transplant | 0.00
  Dissecting Aortic Aneurysm | 0.07
  Diabetic Retinopathy | 0.07
  New-Onset Diabetes | 4.51
  Primary MACE | 4.11
  Primary MACE 2 | 5.77
  Renal Events | 0.07

6. Secondary Outcome: Incidence of Cerebrovascular/Cardiovascular Events Affected by Underlying Risk Factors of Obesity + Blood Glucose Abnormalities + Lipid Abnormalities
Description: Participants reporting cerebrovascular/cardiovascular events who had obesity, blood glucose and lipid abnormalities associated with Blopress at the time of enrollment were reported. The composite events classified under primary MACE1 and primary MACE2 were defined as: MACE1: sudden death, cerebral hemorrhage, cerebral infarction, subarachnoid hemorrhage, and acute myocardial infarction; MACE2: MACE1 + hospitalization for cardiac failure and intervention/hospitalization for angina pectoris. Renal events include (transition to dialysis + renal transplant).
Time Frame: Baseline up to 3 years
Population: as for outcome 3
Measure: Number; unit: Number of events/1,000 person-years
Arm/Group | Candesartan Cilexetil
Number analyzed (Participants) | 3582
Number of events/1,000 person-years
  Sudden Death | 0.35
  Cerebral Hemorrhage | 0.81
  Cerebral Infarction | 3.48
  Subarachnoid Hemorrhage | 0.23
  Acute Myocardial Infarction | 1.28
  Hospitalization for Heart Failure | 0.35
  Intervention/Hospitalization for Angina Pectoris | 2.78
  Atrial Fibrillation | 1.97
  Transition to Dialysis | 0.70
  Renal Transplant | 0.00
  Dissecting Aortic Aneurysm | 0.12
  Diabetic Retinopathy | 0.35
  New-Onset Diabetes | 5.22
  Primary MACE | 6.14
  Primary MACE 2 | 9.27
  Renal Events | 0.70

ADVERSE EVENTS:
Time Frame: Baseline up to 3 years
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Candesartan Cilexetil
Serious Adverse Events (participants affected / at risk) | 320/13804
Other Adverse Events (participants affected / at risk) | 230/13804
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Candesartan Cilexetil (N=13804)
Anaemia (Blood and lymphatic system disorders) | 2
Aplastic anaemia (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 32
Angina pectoris (Cardiac disorders) | 53
Atrial fibrillation (Cardiac disorders) | 7
Atrial flutter (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 9
Cardio-respiratory arrest (Cardiac disorders) | 1
Sick sinus syndrome (Cardiac disorders) | 1
Meniere's disease (Ear and labyrinth disorders) | 1
Goitre (Endocrine disorders) | 1
Blindness unilateral (Eye disorders) | 1
Diabetic retinopathy (Eye disorders) | 1
Retinal artery occlusion (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 2
Small intestinal haemorrhage (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Multi-organ failure (General disorders) | 1
Oedema (General disorders) | 1
Sudden death (General disorders) | 8
Non-cardiac chest pain (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 2
Hepatic ischaemia (Hepatobiliary disorders) | 1
Anaphylactic shock (Immune system disorders) | 1
Cellulitis (Infections and infestations) | 2
Cholangitis suppurative (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Sepsis (Infections and infestations) | 2
Accident (Injury, poisoning and procedural complications) | 1
Cerebral haemorrhage traumatic (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 3
Pneumoconiosis (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 5
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Stress fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood creatinine abnormal (Investigations) | 1
Blood creatinine increased (Investigations) | 5
Blood glucose decreased (Investigations) | 1
Blood glucose increased (Investigations) | 3
Blood potassium increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Glucose urine present (Investigations) | 1
Glycosylated haemoglobin increased (Investigations) | 3
Haemoglobin decreased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Marasmus (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Collagen disorder (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Renal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 20
Cerebral infarction (Nervous system disorders) | 61
Dementia (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Mental impairment (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 4
Transient ischaemic attack (Nervous system disorders) | 4
Completed suicide (Psychiatric disorders) | 1
Azotaemia (Renal and urinary disorders) | 2
Calculus urinary (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Post streptococcal glomerulonephritis (Renal and urinary disorders) | 1
Renal artery stenosis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 10
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1
Spinal operation (Surgical and medical procedures) | 1
Cataract operation (Surgical and medical procedures) | 1
Aortic aneurysm (Vascular disorders) | 1
Aortic dissection (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Iliac artery stenosis (Vascular disorders) | 1
Arteriosclerosis obliterans (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Candesartan Cilexetil (N=13804)
Acute myocardial infarction (Cardiac disorders) | 3
Angina pectoris (Cardiac disorders) | 5
Arrhythmia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 7
Bradycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 4
Sick sinus syndrome (Cardiac disorders) | 1
Supraventricular extrasystoles (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Diabetic retinopathy (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Epigastric discomfort (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest discomfort (General disorders) | 1
Face oedema (General disorders) | 2
Feeling abnormal (General disorders) | 2
Feeling hot (General disorders) | 1
Malaise (General disorders) | 1
Oedema (General disorders) | 2
Oedema peripheral (General disorders) | 2
Thirst (General disorders) | 1
Jaundice (Hepatobiliary disorders) | 2
Liver disorder (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 1
Cholangitis suppurative (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 13
Aspartate aminotransferase increased (Investigations) | 8
Blood cholesterol increased (Investigations) | 5
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 17
Blood glucose increased (Investigations) | 2
Blood potassium increased (Investigations) | 9
Blood pressure abnormal (Investigations) | 1
Blood pressure decreased (Investigations) | 5
Blood triglycerides increased (Investigations) | 8
Blood urea increased (Investigations) | 1
Blood uric acid increased (Investigations) | 16
Gamma-glutamyltransferase increased (Investigations) | 3
Glucose urine present (Investigations) | 2
Glycosylated haemoglobin increased (Investigations) | 3
High density lipoprotein decreased (Investigations) | 2
Low density lipoprotein increased (Investigations) | 1
Weight decreased (Investigations) | 1
Protein urine present (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 7
Gout (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 5
Cerebral infarction (Nervous system disorders) | 5
Depressed level of consciousness (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 25
Dizziness postural (Nervous system disorders) | 5
Headache (Nervous system disorders) | 9
Hypoaesthesia (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 1
Azotaemia (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 3
Erectile dysfunction (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 4
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 3
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 4
Skin discomfort (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3
Photodermatosis (Skin and subcutaneous tissue disorders) | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Orthostatic hypotension (Vascular disorders) | 2
Blood pressure inadequately controlled (Vascular disorders) | 1
Hot flush (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.